CLINICAL TRIAL: NCT01907438
Title: Identification of the Transformation Potential of Normal Estrogen Exposed BRCA1 (Breast Cancer Susceptibility Gene 1) and BRCA2 (Breast Cancer Susceptibility Gene 2) Heterozygous Epithelial Breast Cells Due to Irradiation
Brief Title: Transformation Potential of E2 Exposed Breast Cancer Susceptibility Gene Mutation Heterozygous Epithelial Breast Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Asher Salmon, Asher Salmon, Hadassah Medical Organization
Other Study IDs: ISF-1702/12
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation
Keywords: BRCA; estrogen; epithelial breast cells; genome profile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- non-carriers: Tissues from premenopausal women undergoing esthetic breast surgery with no family history of breast or ovarian cancers will be obtained.epithelial breast cells will be isolated, treated with estrogen for 48 h and then will be irradiated.
- BRCA1 mutation carriers: Tissues from risk-reducing mastectomy in healthy premenopausal women with BRCA1 mutations undergoing.epithelial breast cells will be isolated, treated with estrogen for 48 h and then will be irradiated.
- BRCA2 mutation carriers: Tissues from risk-reducing mastectomy in healthy premenopausal women with BRCA2 mutations undergoing.epithelial breast cells will be isolated, treated with estrogen for 48 h and then will be irradiated.

SUMMARY:
Susceptibility to breast cancer is related to the combination of genetic, hormonal and multiple other environmental risk factors, such as mutations in the BRCA gene and excess exposure to exogenous estrogen, respectively. BRCA is a nuclear protein that maintains genome stability, by acting as a key player in the DNA repair complex. Recently, evidence has emerged that BRCA mutation heterozygosis itself enhances aborted DNA repair and can contribute to breast cancer initiation after exposure to irradiation. In our preliminary results on short-term lymphocyte cultures, we found additional evidence that healthy heterozygous BRCA1 and BRCA2 mutation carriers have a different response to DNA damage than do non-carriers.

The main aim of our ongoing project is to identify the transcriptional modulation and transformation potential of normal BRCA1 and BRCA2 mutation heterozygous epithelial breast cells following irradiation and to examine how it is affected by exposure to estrogen. Our hypotheses will be investigated by RNA-seq and microRNA-seq in order to identify a unique molecular expression profile of the estrogen exposed cells following ionizing irradiation.

Understanding the role of BRCA heterozygosity in cell response to exposure to estrogen and to irradiation may facilitate the development of more appropriate diagnostic and therapeutic strategies for these individuals.

DETAILED DESCRIPTION:
To study the different cell lineages, we plan to isolate and propagate luminal progenitors from a normal human breast tissue. To this end, 10 human breast tissue samples will be obtained from risk-reducing mastectomy in healthy premenopausal women with BRCA1 mutations. Tissues from 10 premenopausal women undergoing esthetic breast surgery with no family history of breast or ovarian cancers will serve as a control group. In order to isolate primary epithelial cells, human mammary tissue will be minced and enzymatically digested overnight in collagenase and hyaluronidase to yield suspension of epithelial organoids. These organoids will be collected and further digested with trypsin, dispase and deoxyribonuclease 1 (DNAse), will be filtered to generate a single cell suspension, resuspended in Hank's + 2% fetal bovine serum (FBS) and 0.1 mg/mL DNAse, and also incubated with a blocking antibody for 15 minutes on ice.

Cells will be treated with estrogen (E2) (10 nM) for 48 h and then will be irradiated for inducing double-strand break. Cells will be irradiated with 8 Gray (Gy) using a Co60 source.

To accomplish our study, estrogen exposed and unexposed BRCA mutation heterozygous epithelial breast cells will be irradiated and 1 h later RNA will be extracted from the cells using Tri-reagent (Sigma). The RNA will be converted to a library of cDNA (complementary DNA) fragments and will be sent for deep sequencing in the illumina Hi-Seq platform.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* premenopausal
* women
* BRCA1 mutations
* BRCA2 mutations

Exclusion Criteria:

* women with breast or ovarian cancer

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: human breast tissue samples will be obtained from risk-reducing mastectomy in healthy premenopausal women with BRCA1 and BRCA2 mutations. Tissues from premenopausal women undergoing esthetic breast surgery with no family history of breast or ovarian cancers also will be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
The transcriptional profile of heterozygous epithelial breast cells | human breast tissue samples will be obtained from premenopausal women undergoing breast surgery. cells will be isolated immediatly and 48h later the transcriptional profile will be identified.
  we will perform a RNA-seq expression profiling analysis of normal estrogen exposed BRCA heterozygous epithelial cells following irradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Y Salmon, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah medical center, Jerusalem, Israel